CLINICAL TRIAL: NCT03222687
Title: Off-label Use of Tacrolimus in Children With Henoch-Schönlein Purpura Nephritis: Effectiveness and Safety
Brief Title: Tacrolimus in Children With Henoch-Schönlein Purpura Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Wei Zhao, Head of department of clinical pharmacy and pharmacology, Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017TAC001
Record Dates: First submitted 2017-07-07; First posted 2017-07-19 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Henoch-Schönlein Purpura Nephritis
Keywords: tacrolimus, Henoch-Schönlein purpura nephritis, children
MeSH Terms: interventions — Tacrolimus; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- therapy group (Experimental): Immunosuppressive therapy included tacrolimus and prednisone.
  Interventions: Drug: tacrolimus; Drug: prednisone

INTERVENTIONS:
Drug: tacrolimus — Immunosuppressive therapy included tacrolimus and prednisone. Tacrolimus treatment was initiated at a dosage of 0.05-0.1 mg/kg/day twice daily and used for at least 6 month. Prednisone was started at 2 mg/kg/day and tapered off gradually after initiation of treatment.
Drug: prednisone — Immunosuppressive therapy included tacrolimus and prednisone. Tacrolimus treatment was initiated at a dosage of 0.05-0.1 mg/kg/day twice daily and used for at least 6 month. Prednisone was started at 2 mg/kg/day and tapered off gradually after initiation of treatment.

SUMMARY:
Henoch-Schönlein purpura (HSP) is the most common vasculitis in children, with an incidence of approximately 10:100 000 children and a slight male predominance (male-to-female ratio of 1.5:1). Henoch-Schönlein purpura nephritis (HSPN) is the principal cause of morbidity for HSP and 1%-7% of HSPN patients may progress to renal failure or end-stage renal disease.

Immunosuppressive therapy has become the standard treatment in children with HSPN, however the use of these drugs are still mainly in an off-label manner in clinical practice. Tacrolimus, a calcineurin inhibitor, has been recently suggested in the treatment of HSPN in children. However, the evidence-based clinical data are still limited.

Given the potential benefits and unmet need in clinical practice, the purposes of this pilot study were to assess effectiveness and safety of tacrolimus in HSPN children and evaluate the potential impact of CYP3A5.

ELIGIBILITY:
Inclusion Criteria:

HSPN children Aged less than 18 years; receiving tacrolimus as initial immunosuppressive therapy -

Exclusion Criteria:

Children received other immunosuppressive drug before the trial or other systemic trial drug therapy; Children had a concomitant medical condition, whose participation, in the opinion of the Investigator and/or medical advisor, may create an unacceptable additional risk.

-

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Complete remission | within 6 months
  clinical symptoms and signs disappeared and proteinuria was less than 4mg/h per m2 body surface area within 6 months.
Partial remission | within 6 months
  if proteinuria was reduced to 4.1-40mg/h per m2 body surface area within 6 months. A nonresponsive patient was defined if there was no improvement in clinical symptoms or signs 6 months after the therapy of tacrolimus with or without prednisone, or urinary protein remained more than 40mg/h per m2 body surface area.
nonresponsive | within 6 months
  A nonresponsive patient was defined if there was no improvement in clinical symptoms or signs 6 months after the therapy of tacrolimus with or without prednisone, or urinary protein remained more than 40mg/h per m2 body surface area.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, Principal Investigator — Shandong University

IPD SHARING:
Plan to Share IPD: No